CLINICAL TRIAL: NCT00000240
Title: Combined Buprenorphine and Behavioral Treatment Without Contingent Reinforcement
Brief Title: Combined Buprenorphine and Behavioral Treatment With and Without Contingent Reinforcement on Opioid and Cocaine Abstinence. - 22
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NIDA-06969-22; R01DA006969 (NIH); R01-06969-22
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 1999-04

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to test combined buprenorphine and behavioral treatment with and without contingent reinforcement on opioid and cocaine abstinence.

ELIGIBILITY:
Please contact site for information.

Ages: 23 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1999-04

PRIMARY OUTCOMES:
Drug use
Retention
Weeks abstinent
Weeks continuous abstinence
Overall treatment outcome
Opioid dependence and psychiatric status

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States